CLINICAL TRIAL: NCT01584180
Title: iCOOL 3 (Induction of COOLing 3): A Randomized Trial Comparing 2 Methods for Rapid Induction of Cooling in Stroke Patients, Cold Infusions vs. EMCOOLS Brain.Pad
Brief Title: A Randomized Trial Comparing 2 Methods for Rapid Induction of Cooling in Stroke Patients, Cold Infusions vs. EMCOOLS Brain.Pad (iCOOL 3)
Acronym: iCOOL 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Sven Poli, Dr. Sven Poli, Consultant Neurologist, Principial Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iCOOL 3
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: hypothermia; induction of hypothermia; cold infusion; local neck cooling; external cooling; surface cooling; non invasive cooling; stroke; intracranial hemorrhage; cerebrovascular disease; neuro intensive care
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Hypothermia; Stroke; Intracranial Hemorrhages; Cerebrovascular Disorders | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold infusions (Active Comparator): Infusion of 1L cold crystalloid solution (4°C) over 15 minutes
  Interventions: Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's
- EMCOOLS Brain.Pad (Active Comparator): Passive external neck cooling with 1 EMCOOLS Brain.Pad (Emergency Medical Cooling Systems AG, Wien, Austria)
  Interventions: Device: EMCOOLS Brain.Pad

INTERVENTIONS:
Drug: Cold crystalloid infusions, 0.9%NaCl or Ringer's — Infusion of max. 1L cold crystalloid solution (4°C) over 15 minutes
  Arms: Cold infusions
Device: EMCOOLS Brain.Pad — Passive external neck cooling with 1 EMCOOLS Brain.Pad
  Other Names: Emergency Medical Cooling Systems AG, Wien, Austria
  Arms: EMCOOLS Brain.Pad

SUMMARY:
Mild hypothermia improves outcome in patients with global cerebral ischemia after cardiac arrest. Hypothermia seems promising also in other acute hypoxic-ischemic or in brain swelling associated cerebrovascular disease. The narrow-time-frame is a major issue ("time is brain"). To provide immediate cooling without delay, easy to use, mobile and effective methods are needed. Cold infusions (4 °C) are an accepted standard worldwide. EMCOOLS Brain.Pad (Emergency Medical Cooling Systems AG, Wien, Austria) is a new non-invasive surface cooling system. A comparison of these two induction methods has never been done before. Neither was the effect of the EMCOOLS Brain.Pad on brain-temperature measured. For the first time iCOOL 3 compares feasibility, safety and efficacy of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Sedation
* Combined ICP-temperature-probe
* Indication to lower body temperature ≤ 1.5°C
* Age ≥ 18 years

Exclusion Criteria:

* Body weight > 120 kg
* Severe renal insufficiency
* Acute pulmonary embolism
* Acute myocardial infarction
* High-grade heart valve stenosis or insufficiency
* Severe cardiac insufficiency (NYHA ≥ III)
* Threatening ventricular dysrhythmia
* Cardiac dysrhythmia with bradycardia (heart rate < 45 /min, QTc > 450 ms, sick sinus syndrome, AV-block II-III°).
* Known hematologic disease with increased risk of thrombosis (e.g. cryoglobulinemia, cold agglutinins, sickle cell anemia)
* Known vasospastic vascular disorder (e.g. Raynaud's phenomenon or thromboangiitis obliterans)
* Skin lesions not allowing a secure application of the EMCOOLS Brain.Pad

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Brain temperature | -15 to +60min
  Primary endpoint: Change of brain temperature during one hour after start of cooling. Repeated measurement ANOVA for within subject contrasts (phase 1 (0 to 15min), 2 (15 to 30min), 3 (30 to 45min) and 4 (45 to 60min)) vs. baseline (-15 to 0min)

SECONDARY OUTCOMES:
(Neuro-)vital parameters | -15 to +180 min
  Effects on (neuro-)vital parameters (e.g. HR, AP, ICP, CPP) are registered
Cerebral autoregulation | 15 to +180 min
  Cerebral auto-regulation parameters (e.g. PRx) are calculated on the basis of the (neuro-)vital parameters monitored.
Safety | 0 - 7 days
  Various safety parameters, such as bleeding complications, cardiac decompensation, or local skin irritations are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Neuro Intensive Care Unit 2, Dept. of Neurology, University Hospital Heidelberg, Heidelberg, Germany